CLINICAL TRIAL: NCT01102010
Title: Postoperative Blood Transfusion for Frail Elderly With Hip Fracture - a Clinical Randomized Controlled Trial
Brief Title: Postoperative Blood Transfusion for Frail Elderly With Hip Fracture
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PBTFEHF
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2013-08

CONDITIONS: Hip Fracture
Keywords: Blood transfusion; Hip fracture; Elderly; Geriatrics; Hospitalization; Frail elderly
MeSH Terms: conditions — Hip Fractures | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood transfusion (Experimental): Restrictive strategy: Blood transfusion when hemoglobin is less than 6 mmol/l (9.7 g/dl)
  Liberal strategy: Blood transfusion when hemoglobin is less than 7 mmol/l (11.3 g/dl)
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — An expanded indication for blood transfusion in the frail elderly

SUMMARY:
Elderly with hip fractures are often frail and discharged from hospital after few days of hospitalisation. Hip fracture surgery is often associated with blood loss, where the patient is at risk of developing anaemia. Low haemoglobin level reduces the body's oxygen transport which causes impaired functional ability and strain on vital organs. Acute anaemia is worse tolerated in elderly, than in younger patients. Therefore this study aims to investigate whether there are effects of an expanded indication for blood transfusion in the frail elderly.

DETAILED DESCRIPTION:
All elderly patients aged 65 and above who are hospitalised from nursing home or sheltered housing facilities to the Orthopaedic Surgery Ward at Aarhus University Hospital with hip fracture and treated operatively, are eligible for this study. According to sample size calculations 284 patients are needed. Informed consent or deputy informed consent, if the patient is cognitively impaired, is needed. Inclusion is dependent on a haemoglobin measure between 6 and 7 mmol/l 6 days after surgery at the latest. Randomization will be computerised. Randomization will determine intervention with blood transfusion and the measurement of haemoglobin is blinded to the patient, relatives, and endpoint assessor. Both transfusion groups will receive blood when haemoglobin is less than 6 mmol/l, as recommended by the Danish Health and Medicine Authority. Geriatric and Orthopaedic Team (GO-team), consisting of following trained specialists: physiotherapist, nurse, and physician, will conduct medical evaluations, including blood transfusions, from admission until 30 days after surgery. The GO-team will work on weekdays both at the Orthopaedic surgery ward and in the patients home immediately after discharge. In accordance with Aarhus Blood Bank's instructions, blood transfusions are given both under hospitalisation, in the nursing homes and in the sheltered housings. Outcomes are functional ability and mortality during 90 days, and overall quality of life (OQoL) after 30 days and 1 year. The association between physical recovery and OQoL are tested.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hip fracture
* Surgery treatment
* Living in nursing homes or sheltered housing facilities
* Haemoglobin level between 6 and 7 mmol/l latest 6th day after surgery
* Written consent

Exclusion Criteria:

* Active cancer
* Pathological fracture
* The patient is against blood transfusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 284 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Functional ability | Measured 10 days after surgery + repeated measurement during 90 days after surgery
  Measurement by Cumulated Ambulation Score (CAS), New Mobility Score (NMS) and Modified Barthel Index (MBI)

SECONDARY OUTCOMES:
Mortality | Measured 30 and 90 days after surgery
  Measurement by the Danish Central Office of Civil Registration
Quality of Life | Measured 30 days and 1 year after surgery
  Measurement by Depression List (DL)

OTHER OUTCOMES:
Delirium | Percentage of participants with delirium measured 10 days after surgery by the score 'Confusion Assessment Method'
  It is an ancillary study to the trial to examine delirium as an outcome in a subsample of 179 nursing home residents. Furthermore, we evaluate if delirium is associated with mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit, Geriatric Department, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836